CLINICAL TRIAL: NCT00682591
Title: Evaluation of Neurocognitive Performance, Quality of Life, and Emotional State in Drug Substituted Patients (Methadone, Buprenorphine, Suboxone) Under Hepatitis C Therapy (Peginterferon Alfa and Ribavirin)
Brief Title: Evaluation of Neurocognitive Performance in Drug Substituted Patients Under Hepatitis C Therapy
Status: Withdrawn | Type: Observational
Why Stopped: Study had to be withdrawn because financial support was cancelled.
Sponsor: University of Wuerzburg (Other)
Responsible Party: Michael Scheurlen, MD (principal investigator), University of Wuerzburg, Germany
Other Study IDs: P05595
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Chronic Hepatitis C Infection
Keywords: hepatitis C; drug substitution; neurocognitive; patients with stable drug substitution therapy; patients with interferon-based antiviral therapy
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Prospective, longitudinal multi-center study performed in 15 participating substitution centers in Germany.

Aims:

- Primary objective: To compare the impact of the different substitution drugs (methadone, buprenorphine, and suboxone) on the neurocognitive, emotional, and quality-of-life-related tolerability in opioid dependent patients under HCV treatment.

- Secondary objective: To investigate if IFN therapy impairs efficacy (with respect to e.g. retention rates, concomitant drug use and in particular neurocognitive function) and tolerability of agonist maintenance treatment with methadone, buprenorphine, or suboxone

ELIGIBILITY:
Inclusion Criteria:

* Opioid-dependent patients on current stable agonist maintenance therapy (for at least 6 months prior to study enrolment) with methadone, buprenorphine, or suboxone.
* Patients need to be infected with chronic hepatitis C and must have indication for therapy with peginterferon alfa and ribavirin.
* Patients with informed written consent with respect to a follow-up of psychiatric side effects and in particular neurocognitive performance.
* Patients with baseline monitoring of emotional state and neurocognitive performance.

Exclusion Criteria:

* According to SPC
* According to legal requirements reg. drug substitution therapy (BTMVV)
* Insufficient knowledge of the German language or cognitive impairment (due to the indispensable application of questionnaires and the TAP, Test Battery of Attentional Performance).
* Age under 18 years or over 65 years
* coinfections such as hepatitis B virus or human immunodeficiency virus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients with chronic hepatitis C infection and drug substitution therapy (methadone, burpenorphine, suboxone)
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2008-07; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Time course of neurocognitive performance (as assessed by the TAP - Test Battery for Attentional Performance) | Repeated measures design with the following evaluation timepoints: baseline, twice to four times during antiviral treatment, twice after antiviral treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Scheurlen, MD, Principal Investigator — Med. Klinik und Poliklinik II, University of Wuerzburg
Locations (1):
- Med. Klinik und Poliklinik II, University of Wuerzburg, Würzburg, Germany

REFERENCES:
- [Background] Kraus MR, Schafer A, Wissmann S, Reimer P, Scheurlen M. Neurocognitive changes in patients with hepatitis C receiving interferon alfa-2b and ribavirin. Clin Pharmacol Ther. 2005 Jan;77(1):90-100. doi: 10.1016/j.clpt.2004.09.007. PMID 15637534
- [Background] Schafer A, Scheurlen M, Weissbrich B, Schottker K, Kraus MR. Sustained virological response in the antiviral therapy of chronic hepatitis C: is there a predictive value of interferon-induced depression? Chemotherapy. 2007;53(4):292-9. doi: 10.1159/000102584. Epub 2007 May 10. PMID 17496415
- [Background] Kraus MR, Schafer A, Faller H, Csef H, Scheurlen M. Psychiatric symptoms in patients with chronic hepatitis C receiving interferon alfa-2b therapy. J Clin Psychiatry. 2003 Jun;64(6):708-14. doi: 10.4088/jcp.v64n0614. PMID 12823087
- [Background] Schafer A, Wittchen HU, Seufert J, Kraus MR. Methodological approaches in the assessment of interferon-alfa-induced depression in patients with chronic hepatitis C - a critical review. Int J Methods Psychiatr Res. 2007;16(4):186-201. doi: 10.1002/mpr.229. PMID 18188838